CLINICAL TRIAL: NCT00253110
Title: A Comparison of Risperidone and Haloperidol for Prevention of Relapse in Subjects With Schizophrenia and Schizoaffective Disorders
Brief Title: A Comparison of Risperidone With Haloperidol in Patients With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006013; RIS-USA-79 (Other: Janssen, LP)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia, Psychotic Disorders; Haloperidol; Risperidone; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Haloperidol

ARMS (2):
- risperidone (Active Comparator)
  Interventions: Drug: risperidone
- haloperidol (Active Comparator)
  Interventions: Drug: haloperidol

INTERVENTIONS:
Drug: risperidone
  Arms: risperidone
Drug: haloperidol
  Arms: haloperidol

SUMMARY:
The purpose of the study is to compare the time to relapse in patients with schizophrenia and schizoaffective disorders receiving risperidone or haloperidol (antipsychotic medications) for at least 1 year.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that causes changes in a person's perception, thoughts, and behaviour. In schizophrenics, the most common symptoms are positive symptoms (delusions and hallucinations), negative symptoms (avoiding social situations, lack of feeling or expression), and disorganized symptoms (confusion in thinking and speech). Schizoaffective disorder is different from schizophrenia, although it may be misdiagnosed as this illness. Schizoaffective disorder is a mental illness distinguished by a combination of a thought disorder (abnormal thinking or psychotic symptoms such as hallucinations or delusions) and a mood disorder (clinical depression or manic component). Manic symptoms include, but are not limited to an overinflated self esteem, increased physical agitation, excessively poor judgment, being easily distracted, and an increased irritability and energy level. This is a randomized, double-blind, parallel-group, controlled study comparing the time to relapse and the incidence of relapse in patients with schizophrenia and schizoaffective disorder being treated with risperidone or haloperidol. The long-term safety and effectiveness of risperidone and haloperidol are also compared. The study is composed of two phases: a 1-week baseline period and a double-blind treatment period. During the baseline period, the doses of risperidone and haloperidol are gradually increased to 4 mg/day for risperidone and 10 mg/day for haloperidol. During the first 4 weeks of double-blind treatment, dosage adjustments can be made in the range of 2 - 8 mg/day for risperidone and 5 - 20 mg/day for haloperidol, based on clinical evaluations of the patient. The double-blind treatment continues at that dose until the last patient entering the study completes 1 year of treatment or for a maximum of 112 weeks. The primary measure of effectiveness is the time to relapse, which is defined using six criteria that indicate the patient's illness is no longer under control (for example, psychiatric hospitalization). Additional efficacy testing conducted includes the Positive and Negative Syndrome Scale for Schizophrenia (PANSS), a rating scale that measures the symptoms of schizophrenia; the Clinical Global Impressions (CGI), a rating system used to evaluate the overall and severity of clinical change in a patient with various diseases affecting the brain; and the Quality of Life Interview (QOLI), a global measure of satisfaction with life. Safety evaluations include the incidence of adverse events, results of clinical laboratory tests (hematology, biochemistry, urinalysis), measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone will be more effective in delaying relapse than haloperidol in patients with schizophrenia and schizoaffective disorder. Risperidone tablets, taken orally, starting at 1 mg/day; increasing to 4 mg/day (Week 1). Haloperidol tablets, taken orally, starting at 2 mg/day; increasing to 10 mg/day (Week 1). After Week 1, dosage may be adjusted (2 - 8 mg/day risperidone; 5 - 20 mg/day haloperidol). Treatment duration >=52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder, according to the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV) criteria
* documented 1-year history of schizophrenia or schizoaffective disorder since the first drug treatment for psychotic symptoms
* history within the previous 24 months of being discharged from an inpatient psychiatric unit, had a partial hospitalization, completed crisis management intervention, or stayed in a hospital emergency room holding area for at least 12 hours
* must have received a stable dose of an antipsychotic medication for the 30 days before study entry
* in the investigator's judgment, must be able to discontinue any current antipsychotic medication.

Exclusion Criteria:

* Patients with clinically significant neurological disorders, with the exception of DSM-IV defined movement disorders that are caused by drugs
* patients with another current DSM-IV Axis I diagnosis (except nicotine or caffeine dependence)
* history or current diagnosis of gastrointestinal, liver, or kidney disease or other condition that might interfere with how the study drug is absorbed, processed, and excreted by the body
* pregnant or nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 1996-05; Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Time to relapse (days)

SECONDARY OUTCOMES:
Change from baseline in total PANSS and PANSS subscale scores and CGI severity score; 1-year relapse rate; QOLI (quality of life); safety evaluations conducted throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- See also: A Comparison of Risperidone with Haloperidol in Patients with Schizophrenia and Schizoaffective Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=349&filename=CR006013_CSR.pdf